CLINICAL TRIAL: NCT05449795
Title: Evaluation of the Performance of Contour Next® and Contour Plus Elite® Blood Glucose Monitoring Systems (BGMS) in Arterial Blood Samples From Hospitalized Adults
Brief Title: Performance of Contour Next® and Contour Plus Elite® BGMS in Arterial Blood Samples From Hospitalized Adults
Status: Completed | Type: Observational
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: GCA-PRO-2021-004-01
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Device: Contour Next and Contour Plus Elite BGMS testing of arterial blood — The purpose of the study is to extend the intended use of two BGMSs to include testing of arterial blood by Health Care Professionals (HCP) in a clinical setting.

SUMMARY:
The purpose of the study is to extend the intended use of two BGMSs to include testing of arterial blood by Health Care Professionals (HCP) in a clinical setting.

DETAILED DESCRIPTION:
This trial will evaluate the performance of both Contour Next BGMS and Contour Plus Elite BGMS using arterial blood from adult patients hospitalized in a Critical Care Unit (medical and surgical intensive care units (ICUs)). The investigational BGMS will be tested by a Point-of-Care (POC) operator in a clinical setting using residual arterial blood samples from adults who underwent prescribed arterial blood tests that were deemed necessary due to their medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years old.
* Residual Arterial blood samples collected from subjects hospitalized in a Critical Care Unit (medical and surgical intensive care units (ICUs)).
* Sample blood volume must be sufficient to complete investigational testing procedures clinical laboratory testing.

Exclusion Criteria:

- Residual arterial blood samples collected from subjects previously enrolled. and evaluated for this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - The subject population will consist of adults who are hospitalized in a Critical Care Unit, (medical and surgical intensive care units (ICUs)) at the Investigational site.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Adelaide Hospital , ICU Research Unit, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: blood samples
Groups:
- Arterial Blood Results: Samples collected and tested in duplicate by BGMS and compared to laboratory results
Period: Overall Study
Arm/Group | Arterial Blood Results
Started | 120; 240 blood samples
Completed | 120; 240 blood samples
Not Completed | 0; 0 blood samples

BASELINE CHARACTERISTICS:
Population: 120 participants were enrolled in the study. Each participant provided two blood samples that were tested. So the number of results analyzed is 240.
Units Other Than Participants: blood samples
Arm/Group | Arterial Blood Results
Number analyzed (Participants) | 120
Number analyzed (blood samples) | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  Australia | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Results From the Contour Next BGMSs Reference Values Within ±12.5% of Reference Values
Description: At least 95% of all blood glucose results shall fall within ±12.5% of reference values (laboratory method) for glucose concentration ≥100 mg/dL(5.55 mmol/L )and within ±12 mg/dL(±0.67 mmol/L) at glucose concentrations <100 mg/dL(5.55 mmol/L).
Time Frame: 1 day
Population: arterial samples
Measure: Count of Units; unit: blood samples
Units Other Than Participants: blood samples
Arm/Group | Arterial Blood Results
Number analyzed (Participants) | 120
Number analyzed (blood samples) | 240
blood samples | 236

2. Primary Outcome: Number of Results From the Contour Plus Elite BGMSs Reference Values Within ±12.5% of Reference Values
Description: At least 98% of values should be within ±12.5% of reference values (laboratory method) for glucose concentration ≥75 mg/dL(4.16 mmol/L) and within ±15 mg/dL(±0.83 mmol/L) at glucose concentrations < 75 mg/dL(4.16 mmol/L).
Time Frame: 1 day
Population: Arterial samples tested.
Measure: Count of Units; unit: blood samples
Units Other Than Participants: blood samples
Arm/Group | Arterial Blood Results
Number analyzed (Participants) | 120
Number analyzed (blood samples) | 240
blood samples | 240

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Arterial Blood Results
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT05449795/Prot_SAP_000.pdf